CLINICAL TRIAL: NCT00426530
Title: A Phase Ib Study Investigating the Combination of Everolimus With Trastuzumab and Vinorelbine in Patients With HER2-overexpressing Metastatic Breast Cancer
Brief Title: Safety of Everolimus in Combination Therapy, in Patients With HER2-overexpressing Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001J2102; 2006-001595-20 (EudraCT Number)
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-04

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: HER2-overexpressing metastatic breast cancer; Breast cancer; Cancer of the breast; Human mammary carcinoma; HER-2; metastatic; everolimus; trastuzumab; vinorelbine
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RAD001 Daily Schedule (Experimental): 5mg or 10mg
  Interventions: Drug: everolimus (RAD001)
- RAD001 Weekly Schedule (Experimental): 30mg
  Interventions: Drug: everolimus (RAD001)

INTERVENTIONS:
Drug: everolimus (RAD001)

SUMMARY:
This study will look at different dose levels and regimens of everolimus combined with weekly trastuzumab and vinorelbine therapy in patients with HER-2 overexpressing metastatic breast cancer.

ELIGIBILITY:
Inclusion criteria:

* Female or male patients ≥18 years with WHO performance status ≤ 1
* HER-2 overexpressing metastatic breast cancer cells confirmed by histology
* Progressive disease on prior trastuzumab alone/or in combination with other anticancer agents, or relapsed any time after completion of this therapy
* Patients neurologically stable with adequate bone marrow, liver and renal function

Exclusion criteria:

* Patients receiving endocrine therapy for breast cancer ≤ 2 weeks prior to study treatment start
* Patients currently receiving chemotherapy, immunotherapy or radiotherapy or who have received these ≤ 4 weeks prior to study treatment start or patients who have received lapatinib ≤ 2 weeks prior to study treatment start
* Patients who have previously received vinorelbine or mTOR inhibitors

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To establish the feasible dose levels/regimens based on End-of-cycle-1 dose limiting toxicity (DLT) | after ever DLT within the first cycle, at least 21 days on treatment, every 2 months from first date of enrollment in a particular regimen

SECONDARY OUTCOMES:
To assess the ability to deliver the trastuzumab and vinorelbine therapy | After LPLV
To assess everolimus, trastuzumab and vinorelbine blood levels in this combination | After LPLV
To evaluate the overall tumor response | every 9 weeks/minus 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (6):
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Stockholm, Sweden

REFERENCES:
- [Derived] Jerusalem G, Fasolo A, Dieras V, Cardoso F, Bergh J, Vittori L, Zhang Y, Massacesi C, Sahmoud T, Gianni L. Phase I trial of oral mTOR inhibitor everolimus in combination with trastuzumab and vinorelbine in pre-treated patients with HER2-overexpressing metastatic breast cancer. Breast Cancer Res Treat. 2011 Jan;125(2):447-55. doi: 10.1007/s10549-010-1260-x. Epub 2010 Nov 25. PMID 21107682
- See also: Results for CRAD001J2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5725